CLINICAL TRIAL: NCT07064057
Title: Effects of Aerobic Training With and Without Sniff Maneuver on Dyspnea, Functional Capacity and Quality of Life Among Asthma Patients
Brief Title: Effects of Aerobic Training With and Without Sniff Maneuver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0341
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Exercise; Dyspnea; Sniff maneuver; Functional capacity; Quality of life
MeSH Terms: conditions — Asthma; Motor Activity; Dyspnea | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercises along with sniff maneuver (Experimental): Aerobic exercises on a stationary bike or electric treadmill three times a week for six weeks.
  Interventions: Other: Aerobic exercise combined with the sniff maneuver technique
- Aerobic exercises only (Active Comparator): The treadmill was used for both the warm-up and cooling-down phases.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise combined with the sniff maneuver technique — Aerobic exercises on a stationary bike or electric treadmill three times a week for six week. Five minutes of stretching, concentrated on the main lower limb muscle groups, were followed by a ten-minute warm-up, twenty minutes of training during the first two weeks and thirty minutes during the third to sixth week, and finally, a five-minute cooling-down phase..
  Arms: Aerobic exercises along with sniff maneuver
Other: Aerobic exercise — The treadmill was used for both the warm-up and cooling-down phases. Heart rate was kept between 40% and 50% of maximum heart rate for these sessions. (5) To achieve a moderate exertion (rated as 11--13 on the Borg scale) and/or a moderate dyspnea (rated as 3---4 on the modified Borg scale), the intensity of the aerobic training was progressively increased.
  Arms: Aerobic exercises only

SUMMARY:
This study was planned to assess effects of Aerobic training with and without Sniff maneuver on Dyspnea, Functional capacity and Quality of life among Asthma Patients. Results showed that when aerobic training done along with the sniff maneuver had proven to be the more effective choice of treatment in reducing severity level of asthma along with the decreased perceived dyspnea and improved quality of life and functional capacity.

DETAILED DESCRIPTION:
This study aimed to check the effects of Aerobic training with and without Sniff maneuver on Dyspnea, Functional capacity and Quality of life among Asthma Patients. This research of randomized clinical trial checked the effects of aerobic training with and without sniff maneuver on dyspnea, functional capacity and quality of life among asthma patient. By taking sample of 28 patients through convenience sampling and randomly allocating them to two group A and B out of which A was received Aerobic training with sniff maneuver and group B was received Aerobic training up to the duration of 3 days per week for 6 weeks. Pre and Post training outcomes of functional capacity was measured through 6 min walk test, dyspnea through Borg rating perceived exertion scale and QOL through 5d euro quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 to 50
* Moderate to severe asthma (FE ratio: 50 to 65%, ˂50%)

Exclusion Criteria:

* Patient with Cardiovascular(5)
* Musculosketal disorders (5)
* Smokers were excluded
* Patient with foot drop
* Osteoarthritis
* Low back pain
* Post traumatic history
* Patients who was suffer physical or mental illness were be excluded
* If participant engage another exercise program were be excluded Mild asthma patient

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Euro QOL 5 Dimensional Questionnaire | 6 weeks
  The EQ-5D is the most often used multi attribute utility (MAU) instrument in cost effectiveness evaluations for evaluating health-related quality of life. The descriptive system is made up of five features: mobility, self-care, regular activities, pain/discomfort, and anxiety/depression. The terms "not /no problems," "slight problems," "moderate problems," "severe problems," and "unable to" (mobility, self-care, regular activities) are used to describe the five levels in each category. Other terms used are "extreme" (pain/depression) or "extremely" (anxiety/depression). The patient is questioned to rate his or her current state of health by checking the box next to the statement that most closely matches each of the five dimensions.
Borg Scale | 6 weeks
  Dyspnea was checked by Borg Scale.
6 Min Walk Test | 6 weeks
  Functional capacity was checked by 6 min walk test Stopwatch to calculate overall activity time

CONTACTS AND LOCATIONS:
Overall Officials: Hira Shaukat, Mphill, Principal Investigator — Riphah International University
Locations (1):
- Al-Zahra Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moraes-Ferreira R, Brandao-Rangel MAR, Gibson-Alves TG, Silva-Reis A, Souza-Palmeira VH, Aquino-Santos HC, Frison CR, Oliveira LVF, Albertini R, Vieira RP. Physical Training Reduces Chronic Airway Inflammation and Mediators of Remodeling in Asthma. Oxid Med Cell Longev. 2022 Oct 20;2022:5037553. doi: 10.1155/2022/5037553. eCollection 2022. PMID 36312895
- [Background] Hansen ESH, Pitzner-Fabricius A, Toennesen LL, Rasmusen HK, Hostrup M, Hellsten Y, Backer V, Henriksen M. Effect of aerobic exercise training on asthma in adults: a systematic review and meta-analysis. Eur Respir J. 2020 Jul 30;56(1):2000146. doi: 10.1183/13993003.00146-2020. Print 2020 Jul. PMID 32350100
- [Background] Andrade LB, Britto MC, Lucena-Silva N, Gomes RG, Figueroa JN. The efficacy of aerobic training in improving the inflammatory component of asthmatic children. Randomized trial. Respir Med. 2014 Oct;108(10):1438-45. doi: 10.1016/j.rmed.2014.07.009. Epub 2014 Aug 29. PMID 25231109
- [Background] Abdelbasset WK, Alsubaie SF, Tantawy SA, Abo Elyazed TI, Kamel DM. Evaluating pulmonary function, aerobic capacity, and pediatric quality of life following a 10-week aerobic exercise training in school-aged asthmatics: a randomized controlled trial. Patient Prefer Adherence. 2018 Jun 15;12:1015-1023. doi: 10.2147/PPA.S159622. eCollection 2018. PMID 29942118